CLINICAL TRIAL: NCT03643796
Title: The Effect of a Narcotic Free Total Intravenous Anesthesia on the Outcome and Patient Safety During Anterior Cervical Discectomy and Fusion (ACDF) Surgery: A Randomized Controlled Trial
Brief Title: Narcotic Free TIVA and Incidence of Unacceptable Movements Under Anesthesia During ACDF Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207374
Record Dates: First submitted 2018-07-05; First posted 2018-08-23 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-04

CONDITIONS: Anterior Cervical Discectomy and Fusion (ACDF)
MeSH Terms: interventions — Remifentanil; Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remifentanil Group (Active Comparator): Remifentanil infusion of 0.05 to 0.2 mcg/kg/minute started just prior to induction and stopped at emergence from anesthesia.
  Interventions: Drug: Remifentanil
- Ketamine and Dexmedetomidine group (Active Comparator): dexmedetomidine bolus of 0.5 mcg/kg over 10 minutes starting 5 minutes prior to induction followed by an infusion of 0.2-0.7 mcg/kg/hour that will be stopped with the start of closing the surgical wound.
  Ketamine infusion of 2 mcg/kg/minute will be started at induction. It will be stopped at the beginning of the emergence from anesthesia, roughly 45 minutes from extubation.
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remifentanil — Remifentanil infusion of 0.05 to 0.2 mcg/kg/minute started just prior to induction and stopped at emergence from anesthesia.
  Arms: Remifentanil Group
Drug: Ketamine — Ketamine infusion of 2 mcg/kg/minute will be started at induction. It will be stopped at the beginning of the emergence from anesthesia, roughly 45 minutes from extubation.
  Arms: Ketamine and Dexmedetomidine group
Drug: Dexmedetomidine — dexmedetomidine bolus of 0.5 mcg/kg over 10 minutes starting 5 minutes prior to induction followed by an infusion of 0.2-0.7 mcg/kg/hour that will be stopped with the start of closing the surgical wound.
  Arms: Ketamine and Dexmedetomidine group

SUMMARY:
This study will help the investigators learn more about the best way to give anesthesia for these kinds of surgery. The investigators will be using 2 different groups of medications that is commonly used in ACDF surgery, one group has a Narcotic, and the other group does not. The investigators wish to test whether a narcotic free anesthetic will result in an overall safer surgery, better patient recovery, and satisfaction. The investigators think also that eliminating the Narcotic from the Anesthetic regimen will allow patients to recover faster after surgery , and consume less pain medicines in the postoperative period.

ELIGIBILITY:
Inclusion Criteria

* Men and women 18- to 80-years old
* ASA 1, 2, 3
* 1 or 2 levels ACDF

Exclusion Criteria

* ASA 4
* Seizure disorders
* Chronic narcotic use
* Opiate abuse
* Major cardiac comorbidity, or significantly elevated blood pressure
* Known hypersensitivity to fentanyl analogs, ketamine, or propofol injectable emulsions.
* Known allergy to eggs, egg products, soybeans, or soy products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdeldayem, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was all done in the Preoperative area at the morning of the surgery
Pre-assignment Details: No wash outs or run-in has occurred
Period: Overall Study
Arm/Group | Remifentanil Group | Ketamine and Dexmedetomidine Group
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil Group | Ketamine and Dexmedetomidine Group | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 2 | 3 | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 46 (20) | 52 (19) | 49 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Unacceptable Movement Under General Anesthesia
Description: Gross visible movement reported by the anesthesiologist or surgical team: bucking, chewing, or reaching to the endotracheal tube and induced by nociception, or head manipulation and positioning by the surgical or anesthesiology team or during a motor evoked potential stimulation.
Time Frame: duration of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil Group | Ketamine and Dexmedetomidine Group
Number analyzed (Participants) | 15 | 17
Participants | 1 | 1

2. Secondary Outcome: Hemodynamic Stability
Description: Any increase in the heart rate by more than 20% of patient baseline before induction of anesthesia
Time Frame: up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil Group | Ketamine and Dexmedetomidine Group
Number analyzed (Participants) | 15 | 17
Participants | 4 | 5

3. Secondary Outcome: Time to Extubation
Description: From start of of emergence from anesthesia until time of extubation. Shorter amount of time between the two, is desired.
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Ketamine and Dexmedetomidine Group: dexmedetomidine bolus of 0.5 mcg/kg over 10 minutes starting 5 minutes prior to induction followed by an infusion of 0.2-0.7 mcg/kg/hour that will be stopped with the start of closing the surgical wound.
  Ketamine infusion of 2 mcg/kg/minute will be started at induction. It will be stopped at the beginning of the emergence from anesthesia, roughly 45 minutes from extubation.
  Ketamine: Ketamine infusion of 2 mcg/kg/minute will be started at induction. It will be stopped at the beginning of the emergence from anesthesia, roughly 45 minutes from extubation.
  Dexmedetomidine: dexmedetomidine bolus of 0.5 mcg/kg over 10 minutes starting 5 minutes prior to induction followed by an infusion of 0.2-0.7 mcg/kg/hour that will be stopped with the start of closing the surgical wound.
Arm/Group | Remifentanil Group | Ketamine and Dexmedetomidine Group
Number analyzed (Participants) | 15 | 17
minutes | 12 (7) | 18 (7)

4. Secondary Outcome: Quality of Recovery
Description: ( Modified Quality of Recovery score, QoR-15) is a psychometric assessment of recovery from general anesthesia.Answers of 15 questions are given scores from 1 to 10 on a Likert scale. The score ranges from 0 to 150. The questionnaire is designed to assess the emotional state, physical comfort, psychological support, physical independence, and pain. A higher score indicates a better outcome
Time Frame: 24 hours post-op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine and Dexmedetomidine Group | Remifentanil Group
Number analyzed (Participants) | 17 | 15
units on a scale | 122 (7) | 127 (8)

5. Secondary Outcome: Narcotic Consumption
Description: all narcotics and pain medication consumed by subject in the recovery room until discharged will be recorded and compared among 2 study groups.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Morphine Equivalents
Arm/Group | Remifentanil Group | Ketamine and Dexmedetomidine Group
Number analyzed (Participants) | 15 | 17
Morphine Equivalents | 12.7 (2.4) | 11.5 (2.7)

ADVERSE EVENTS:
Time Frame: 3 years , 9 months
Arm/Group | Ketamine and Dexmedetomidine Group | Remifentanil Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT03643796/Prot_SAP_000.pdf